CLINICAL TRIAL: NCT04110249
Title: A Pilot Study of Photoacoustic Imaging (PAI) in H&Amp;N Cancer Patients
Brief Title: Photoacoustic Imaging for Measuring Tumors and Normal Tissue in Patients With Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: equipment issues
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 48917; NCI-2019-06045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 48917 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); R01CA204636 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-10-01 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Carcinoma; Head and Neck Lymph Node; Head and Neck Squamous Cell Carcinoma; Laryngeal Neoplasm; Radiation Therapy Recipient
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (PAI, ALTENS) (Experimental): PART I: Patients undergo PAI before the start of chemoradiation therapy, weekly during 7 weeks of chemoradiation, and again 3-4 months after completion of chemoradiation therapy.
  PART II (CANCER-FREE WITH XEROSTOMIA): Patients undergo PAI at baseline, up to twice during acupuncture-like transcutaneous nerve stimulation (ALTENS) therapy, once after ALTENS, and at 3-6 months follow up.
  Interventions: Procedure: Photoacoustic Imaging; Procedure: Transcutaneous Acupoint Electrical Stimulation

INTERVENTIONS:
Procedure: Photoacoustic Imaging — Undergo PAI
Procedure: Transcutaneous Acupoint Electrical Stimulation — Undergo ALTENS
  Other Names: acupuncture-like transcutaneous electrical nerve stimulation; ALTENS; TAES

SUMMARY:
This trial studies how well photoacoustic imaging works in measuring tumors and normal tissue in patients with head and neck cancer. Photoacoustic imaging (PAI) is a low-risk imaging method that provides information about the oxygenation of tissues using a combination of light and ultrasound techniques. This study may help doctors determine if PAI is correlated with clinical responses of both tumor (for example: shrinking, swelling or disappearing) and normal tissues (for example: skin redness, dry mouth, appearance of sores, healing of skin or mucosa). If there is a correlation with clinical responses, then doctors may develop PAI as method for measuring response to earlier treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Define the feasibility of the current photoacoustic imaging (PAI) technology in head and neck (H&N) cancer patients.

SECONDARY OBJECTIVE:

I. Define the utility of the current PAI in H&N cancer patients.

OUTLINE:

PART I: Patients undergo PAI before the start of chemoradiation therapy, weekly during 7 weeks of chemoradiation, and again 3-4 months after completion of chemoradiation therapy.

PART II (CANCER-FREE WITH XEROSTOMIA): Patients undergo PAI at baseline, up to twice during acupuncture-like transcutaneous nerve stimulation (ALTENS) therapy, once after ALTENS, and at 3-6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* No restriction on race or ethnic background
* Subject must understand the investigational nature of the study and sign an independent ethics committee/institutional review board approved written informed consent prior to receiving any study related procedure
* FOR CANCER PATIENTS IN THE H&N RADIATION GROUP (PART I):
* Biopsy-confirmed diagnosis of head and neck squamous cell carcinoma (HNSCC) getting chemoradiation therapy
* Presence of neck nodes or laryngeal tumor superficial enough (within 2-3 cm of skin surface) to allow imaging by photoacoustic ultrasound (PA-US)
* FOR ALTENS PATIENTS (PART II):
* History of prior radiation therapy with xerostomia requiring ALTENS

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unwilling or unable to follow protocol requirements or provide consent
* Any condition which in the Investigator?s opinion deems the subject an unsuitable candidate to undergo imaging procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of photoacoustic imaging (PAI) to quantify tumor characteristics (part I): rate | Up to 6 months after treatment completion
  Feasibility rate is defined as the proportion of evaluable patients who have at least 3 imaging sessions that produce a usable image.
Feasibility of PAI to quantify tumor characteristic in patients undergoing ALTENS (part II): rate | Up to 2 years
  Feasibility rate is defined as the proportion of evaluable patients who have at least 3 imaging sessions that produce a usable image.

SECONDARY OUTCOMES:
Utility of serial PAI-based oxygen saturation (%sO2) measurements | Up to 2 years
  Descriptive statistics (means, medium) will be used to summarize percent of SO2
Changes in hemoglobin (hbt) measurements | Up to 2 years
  Compare hemoglobin measurements between baseline until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States